CLINICAL TRIAL: NCT02308436
Title: Prophylactic Effect of a CANDIDA Mouthwash, Containing the Curolox™ Peptide: a Mono-centre, Not-controlled. Not Blinded, Not-randmised in Situ Study
Brief Title: Prophylactic Effect of a CANDIDA Mouthwash, Containing the Curolox™ Peptide
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is not realised.
Sponsor: Mibelle AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P11-4-MW15.042
Record Dates: First submitted 2014-11-27; First posted 2014-12-04 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Erosion of Teeth, Unspecified
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Candida Mouthwash with Curolox™ Peptide (Experimental): Repeated applications 2.5 ml or 5 ml twice daily
  Interventions: Device: Candida Mouthwash with Curolox™ Peptide

INTERVENTIONS:
Device: Candida Mouthwash with Curolox™ Peptide — Prophylaxis - protection and care of teeth against caries & acidic challenges
  Other Names: Candida Protect

SUMMARY:
In vitro results showed a protective effect against acids for the mouthwash containing Curolox™ peptide. The goal of this in situ study is to detect the Curolox™ peptide under natural oral conditions on the tooth surface and to proof the in vitro results obtained. So far there are no effect and safety data of the Curolox™ mouthwash under natural oral conditions available.

DETAILED DESCRIPTION:
The primary objective of the study is the detection of the Curolox™ peptide on the bovine enamel sample (proof-of-concept) under in vivo conditions after rinsing with the peptide-containing mouth wash.

Secondary Objectives

The secondary objectives of the study are:

1. safety and tolerance of the mouthwash in participants
2. identification of the duration the Curolox™ peptide is present on the bovine tooth surface under in vivo conditions
3. identification of the most effective mouthwash rinsing volume (2.5 mL or 5 mL)
4. prophylactic effect of multiple applications of the mouthwash confirmation of the prophylactic effect of the Curolox™ peptide obtained in in vitro study

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and to follow the study procedures and instructions
* Willing to wear a dental appliance for 7 days
* Willing and able to attend the on-study visits
* Good oral hygiene throughout the study
* Written informed consent before participation in the study

Exclusion Criteria:

* Volunteer with an active periodontal disease or periodontal surgery < 1 year prior to study participation
* Volunteer with hypersensitive teeth or with any other (painful) oral pathology or defect
* Volunteer with an orthodontic appliance
* Volunteer undergoing a medical treatment
* Volunteer who is allergic to dental products
* Pregnant and lactating woman
* Concurrent participation in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Detection of Curolox peptide by mass spectroscopy | Immediately after rinsing with the mouthwash
  The primary outcome is the detection of the Curolox™ peptide on the bovine enamel sample immediately after rinsing with the peptide-containing mouth wash by mass spectroscopy

SECONDARY OUTCOMES:
Detection of Curolox peptide by mass spectroscopy | 12 hours, 24 hours, 48 hours, 96 hours
  The secondary outcome is the detection of the Curolox™ peptide on the bovine enamel sample 12 hours, 24 hours, 48 hours and 96 hours after rinsing with the peptide-containing mouth wash by mass spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Christian Besimo, Dr.med.dent., Principal Investigator — Aeskulap Klinik; Ulrich P. Saxer, Dr.med.dent., Study Director — Aeskulap Klinik / PZZN
Locations (1):
- Aeskulap Klinik, Brunnen, Switzerland